CLINICAL TRIAL: NCT06937164
Title: Beliefs and Expectation Effects on Blood Pressure Following Isometric Exercise in Inactive Adults
Brief Title: Blood Pressure Following Isometric Exercise in Inactive Adults
Acronym: BELIEF-BP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Canterbury Christ Church University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: ETH2223-0326
Record Dates: First submitted 2025-04-07; First posted 2025-04-22 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-04

CONDITIONS: Hypertension; Elevated Blood Pressure; Sedentary Lifestlye
Keywords: Isometric Exercise; Blood Pressure; Post-Exercise Hypotension; Physical Inactivity; Heart Rate Variability; Electromyography (EMG); Muscle Fatigue; Cardiovascular Adaptation; Exercise Intervention; Non-Pharmacological Treatment; Hypertension Prevention; Autonomic Nervous System; BELIEF-BP
MeSH Terms: conditions — Hypertension; Post-Exercise Hypotension; Sedentary Behavior

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned to one of three parallel groups: (1) isometric exercise training (IET) with neutral information, (2) IET with expectation-enhancing information, or (3) a no-intervention control group. Intervention groups complete repeated isometric leg extension sessions across multiple visits. Prior to training, participants receive distinct information to influence their beliefs about IET. The control group does not receive training or information. Participants are blinded to group assignment, and outcomes such as blood pressure, heart rate variability, and muscle fatigue are assessed independently across groups.
Who Masked: Participant
Masking Description: Participants are blinded to group assignment. They are not informed whether they are receiving neutral or expectation-enhancing information, or whether they are in a control group. Due to the nature of the study, the researcher is not blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Neutral Information + Isometric Exercise (Experimental): Participants in this group complete repeated isometric exercise training sessions. Prior to training, they receive a neutral informational presentation about isometric exercise, which does not mention blood pressure or cardiovascular benefits. The exercise consists of bilateral isometric leg extensions on a dynamometer. Cardiovascular and neuromuscular outcomes, including blood pressure, heart rate variability, and muscle fatigue, are monitored throughout the intervention period.
  Interventions: Behavioral: Isometric Exercise Training (IET)
- Expectation-Enhancing Info + Isometric Exercise (Experimental): Participants in this group complete repeated isometric exercise training sessions. Prior to training, they receive an expectation-enhancing informational presentation that emphasizes the effectiveness of isometric exercise as a non-pharmacological intervention for reducing blood pressure. The exercise consists of bilateral isometric leg extensions on a dynamometer. Blood pressure, heart rate variability, and muscle activity are assessed to determine physiological responses to the intervention.
  Interventions: Behavioral: Isometric Exercise Training (IET); Behavioral: Expectation-Enhancing Informational Framing
- No-Intervention Control (No Intervention): Participants in this group do not receive any intervention or educational presentation. They attend study visits for assessment purposes only. Measurements include resting blood pressure, heart rate variability, and muscle activity, allowing for comparison with the intervention groups to evaluate the effects of isometric exercise training.

INTERVENTIONS:
Behavioral: Isometric Exercise Training (IET) — Participants perform four repetitions of 90 degree bilateral isometric leg extensions on a dynamometer at 30% of their maximum voluntary contraction (MVC). Each contraction is held for 2 minutes, with 2-minute rest intervals between bouts. Sessions are performed three times per week for four weeks. This behavioral intervention is designed to investigate the acute and chronic effects of isometric exercise on blood pressure, heart rate variability, and muscle fatigue.
  Other Names: Static Strength Training; Leg Extension Hold Training
  Arms: Expectation-Enhancing Info + Isometric Exercise; Neutral Information + Isometric Exercise
Behavioral: Expectation-Enhancing Informational Framing — Participants receive a brief standardized presentation highlighting isometric exercise as an evidence-based intervention for lowering blood pressure. The presentation includes statements designed to enhance outcome expectations based on prior literature and expert framing.
  Arms: Expectation-Enhancing Info + Isometric Exercise

SUMMARY:
This study investigates how isometric exercise training (IET) affects blood pressure in physically inactive adults. Isometric exercise involves sustained muscle contractions without movement-for example, pushing against a fixed object. Previous research has shown that IET may help reduce blood pressure, but the mechanisms involved are not fully understood.

The purpose of this study is to assess both the immediate (acute) and long-term (chronic) effects of IET on cardiovascular outcomes. Participants will complete a series of lab-based exercise sessions over several weeks. In these sessions, they will perform repeated bouts of isometric leg extensions while seated on an exercise machine designed to measure muscle force.

Throughout the study, researchers will monitor participants' blood pressure, heart rate, and muscle activity. Acute responses-such as post-exercise hypotension (a short-term drop in blood pressure)-will be measured immediately after exercise. Chronic changes, such as resting blood pressure improvements, will be evaluated across the training period.

Additional measurements will include heart rate variability (HRV), which gives insight into autonomic nervous system activity, and electromyography (EMG), which tracks muscle fatigue and activation patterns. These data will help explore potential mechanisms behind the cardiovascular benefits of IET.

By examining how repeated sessions of isometric exercise influence blood pressure and related physiological responses, this research may support the use of IET as a non-pharmacological strategy for managing or preventing hypertension in physically inactive individuals.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Self-reported physically inactive or insufficiently active (not meeting current physical activity guidelines)
* Not currently engaged in structured resistance or isometric exercise training
* Able to attend lab sessions over a 4-week period
* Provides written informed consent

Exclusion Criteria:

* Current diagnosis of hypertension requiring medication
* Any known cardiovascular, neurological, or musculoskeletal condition contraindicating isometric exercise
* Formal education or professional background in exercise science, physiology, or a related field
* Pregnant or planning to become pregnant during the study period
* Inability to follow verbal instructions or complete study protocols

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-04-21 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Change in Resting Systolic Blood Pressure | Baseline to Post-Intervention (approximately 4 weeks)
  Systolic blood pressure will be measured at rest using a Task Force Monitor prior to and after the isometric exercise intervention period. The primary outcome is the change in resting systolic blood pressure from baseline to final testing. Measurements are taken in a seated position following standard resting protocols.

SECONDARY OUTCOMES:
Change in Diastolic Blood Pressure | Baseline to Post-Intervention (approximately 4 weeks)
  Diastolic blood pressure will be assessed in the same manner as systolic. The secondary outcome is the change in diastolic values from baseline to final testing.
Post-Exercise Hypotension Response | During the first week of the exercise intervention. Sessions 1, 2 and 3.
  Post-exercise hypotension will be evaluated as the change in systolic and diastolic blood pressure immediately following each isometric exercise session, compared to pre-exercise baseline.
Change in Heart Rate Variability (HRV) | Baseline to Post-Intervention (approximately 4 weeks)
  HRV will be analyzed using Task Force Monitor data to assess autonomic modulation. Measures include time-domain (e.g., RMSSD) and frequency-domain (e.g., LF/HF ratio) indices.
Change in Muscle Fatigue Markers (EMG) | Baseline to Post-Intervention (Approximately 4 weeks)
  Muscle fatigue will be assessed using surface electromyography (EMG) of the vastus lateralis. Fatigue indices include changes in median frequency and torque stability over repeated contractions.

CONTACTS AND LOCATIONS:
Overall Officials: Sean Machak, Principal Investigator — Canterbury Christ Church University
Locations (1):
- Canterbury Christ Church University, Canterbury, Kent, United Kingdom

IPD SHARING:
Plan to Share IPD: No
This is an early-phase investigator-led study involving a small sample size. At this stage, there are no plans to share individual participant data due to ethical and data governance constraints outlined in the approved protocol. Aggregated results may be shared through publication or presentation.